CLINICAL TRIAL: NCT06624527
Title: The Effect of Cognitive Behavior Therapy-Based Psychoeducation Given to Children With Attention Deficit Hyperactivity Disorder on Children's Quality of Life, Anxiety and Depression
Brief Title: Cognitive Behavior Therapy for Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Vedat ARGIN, Lecturer, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VA_001; 323S282 (Other Grant/Funding Number: Scientific and Technical Research Council of Turkey)
Record Dates: First submitted 2024-09-26; First posted 2024-10-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Child,; Attention deficit Hyperactivity disorder; Cognitive Behavioral Therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This study was planned as a pre-test/post-test, single blind randomized controlled experimental design
Who Masked: Participant
Masking Description: In this study, the sample group was determined in the masking process. The sample group was divided into a control group and an intervention group using a random sampling method. It was not disclosed which group the participants were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention will be made to the control group. This group will be given a first test using the scales specified in the data collection, and a final test will be given 30 days later using the same scales.
- Intervention group (Experimental): After the first test application with the scales specified in the data collection, 8 sessions of Cognitive Behavior Therapy-based psycho-education sessions will be applied to the intervention group. At the end of the 8 sessions (which will last 30 days on average), a final test will be applied.
  Interventions: Other: Psychoeducation based on Cognitive Behavioral Therapy

INTERVENTIONS:
Other: Psychoeducation based on Cognitive Behavioral Therapy — A psycho-educational application based on Cognitive Behavior Therapy consisting of a total of 8 sessions prepared by the researcher.
  Arms: Intervention group

SUMMARY:
The aim of this study was planned to determine the changes that cognitive behavior therapy-based psycho-education against the negativities brought by the disease in the long term of children diagnosed with Attention Deficit Hyperactivity Disorder will create changes in the child's quality of life, anxiety and depression status and disease symptoms.

As a result of this study, if cognitive behavior-based psycho-education has a positive effect on anxiety, depression and quality of life of children with Attention Deficit Hyperactivity Disorder, it is thought to contribute positively to the development of the disease for the sick child and parents by organizing psycho-education programs with the training to be given to child health nurses.

DETAILED DESCRIPTION:
1. Research Model This study was planned as a pre-test/post-test, single blind randomized controlled experimental design.
2. Hypotheses of the Study Hypothesis 1 (H1): Does cognitive behavior therapy-based psycho-education given to children with ADHD affect children's quality of life? Hypothesis 2 (H2): Does cognitive behavior therapy-based psycho-education given to children with ADHD affect children's anxiety and depression levels?
3. Place and Time of the Study This study was conducted at Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital / Department of Child and Adolescent Psychiatry between September 25, 2023 and December 30, 2024.
4. Ethical Aspects of the Study

   * With the decision numbered 2022/29 of Hasan Kalyoncu University Health Sciences Institute Board of Directors, this research was accepted as a doctoral thesis subject on 19.12.2022.
   * Ethics committee permission was obtained from Hasan Kalyoncu University Faculty of Health Sciences Non-Interventional Research Ethics Committee with the decision numbered 2023/31 dated 31.01.2023.
   * Written institutional permission was obtained from Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital, where the research will be conducted, with decision number 24523 dated 22.09.2023.
   * Within the scope of the research, "CBT Practitioner Training in Children and Adolescents" was received from Fatih Sultan Mehmet University (Barcode No: UN_041054323475554869027).
   * The research was supported by the Scientific and Technical Research Council of Turkey 1002- A Rapid Support (Project No: 323S232).
   * For the scales used in the study, permission was obtained from the scale developers via e-mail.
   * Within the scope of the study, all participants who agreed to participate in the study were given preliminary information about the study.
   * Confidentiality of patients' names and information was taken as a basis.
   * No fee was requested from the patients to participate in the study and no additional payment was made to the patients participating in the study.
   * Participation in the study was voluntary.
5. Population and Sample of the Study The population of the study consisted of all children with ADHD (newly diagnosed children and children who were followed up) and their parents who applied to the outpatient clinic.

   The sample of the study consisted of patients who met the inclusion criteria and agreed to participate in the study. Before starting the study to determine the sample size, reference results were evaluated based on literature reviews. In line with the data entered into the G Power 3.1.9.7 program, alpha: 0.05, effect size 0.8, confidence interval 95%, the number of participants to be included in the study for each group was calculated as at least 35 children and 35 parents for the control and intervention groups separately, for a total of 70 control and 70 intervention groups. Considering the losses during the study, the study was started with groups of 40 participants each.
6. Sample Inclusion Criteria Criteria for children's participation in the study;

   * Diagnosed with ADHD according to DSM-V diagnostic criteria,
   * No other comorbid disease accompanying ADHD,
   * No mental disability,
   * Not receiving pharmacological treatment,
   * 8-16 years old,
   * Can read and write,
   * Communication and cooperation,
   * Children who agree to participate in the study (their parents and/or themselves) will be included in the study.

   Criteria for parental participation in the study:
   * Allowing their child to participate in the study,
   * Living with her child,
   * the child's natural parent,
   * No hearing-speech impairment,
   * Without a diagnosed and treated mental illness,
   * Mothers who can communicate and are open to cooperation will be included in the study.
7. Data Collection Tools In the collection of data, the "Personal Information Form" created in line with the literature, the "Revised Children's Anxiety and Depression Scale" filled out separately by the child and the parent to determine the anxiety and depression levels of children, and the "Quality of Life Scale for Children" to determine the quality of life of children were used.

   7.1 Descriptive Characteristics Form The "Personal Information Form" prepared by the researcher included 6 questions for the child/adolescent and 14 questions for the parents to determine the sociodemographic variables (age, gender, education level, occupation, marital status, monthly income, school achievement) and information about the disease.

   7.2 Quality of Life Scale in Children It is a scale developed by Varni et al. in 1999 as a result of a 15-year study to measure the physical and psychosocial experiences of children between the ages of 2-18, independent of illness, and their health-related quality of life. Physical health, emotional and social functioning areas and school functioning areas, which are the characteristics of the state of health defined by the World Health Organization, are questioned in the scale. The scale consists of 23 items in total and is prepared as a four-point Likert scale. In the reliability assessment of the scale, Cronbach's alpha coefficient was found to be 0.93. Item scores are evaluated between 0 and 100. If the answer to the question is marked as never, it gets 100 points. If it is marked as "rarely" it gets 75 points, if it is marked as "sometimes" it gets 50 points, if it is marked as "frequently" it gets 25 points and if it is marked as "almost always" it gets 0 points. A person's health-related quality of life is considered to be more positive the higher the total score.

   Scale scoring is carried out in three different areas; Scale Total Score (SCS), Physical Health Total Score (PHTS) and Psychosocial Health Total Score (PSTP), which assess emotional, social and school functioning.

   The validity and reliability study of the scale in Turkish was conducted by Üneri for 2-7 age groups and Çakın Memik for 8-18 age groups. Internal consistency study was conducted for reliability assessment and Cronbach's alpha coefficient was found to be 0.93. Validity assessment was made by looking at construct validity and clinical validity. In this study, Cronbach's alpha coefficient was found to be 0.94.

   7.3. Anxiety and Depression Scale in Children-Child/Parent Form The Revised Anxiety and Depression Scale (RADS) is a clinical symptom screening scale developed to detect DSM-IV based depression and anxiety disorders in children and adolescents.

   It was developed by Chorpita et al. in 2000 and has a parent and child form that can be completed independently. Consisting of 47 items, the child and parent scale forms consist of 6 sub-dimensions in total.

   These dimensions are Separation Anxiety (items 5, 9, 17, 18, 33, 45, 46), Social Phobia (items 4, 7, 8, 12, 20, 30, 32, 38, 43), Obsessive Compulsive Disorder (items 10, 16, 23, 31, 42, 44), Panic Disorder (items 3,14,24,26,28,34,36,39,41. items), Generalized Anxiety Disorder (items 1,13,22,27,35,37) and Major Depressive Disorder (items 2,6,11,15,19,21,25,29,40,47). In the scale score calculation; a total of eight scores can be calculated. These scores represent the total scores of the scale, also known as the six sub-dimensions, anxiety total score and anxiety-depression total score.

   To calculate the total anxiety score, items for social phobia, panic disorder, separation anxiety disorder, generalized anxiety disorder and obsessive-compulsive disorder are summed. For the total anxiety-depression score, the major depressive disorder score is added.

   The Cronbach's alpha coefficients of the sub-dimensions in the original form of the scale are as follows: 0.82 for Social Phobia, 0.79 for Panic Disorder, 0.76 for Separation Anxiety Disorder, 0.76 for Major Depressive Disorder, 0.73 for Obsessive Compulsive Disorder and 0.77 for Generalized Anxiety Disorder.

   In the study conducted by Görmez et al. in 2017, the scale was adapted to Turkish and validity and reliability studies were conducted. The Turkish version of the scale consists of 47 items and has a four-point Likert scale (0=never, 1=sometimes, 2=often and 3=always).

   The six-factor sub-dimensions of the scale were confirmed by confirmatory factor analysis and the internal consistency of the Turkish form was strong/excellent with a Cronbach alpha score of .95. The sub-dimensions ranged from .75 to .86. There is sufficient evidence to prove that it is a valid scale for use with Turkish children and adolescents. In this study, Cronbach's alpha coefficient was 0.92.

   After the child and parent scales are completed, the child's gender and age are recorded in the scoring table and T and Raw scores are determined. RCADS-Parent: scoring was done using the Excel program version 32. Any sub or total scale T score, scores of 65 and above indicate borderline clinical threshold, while scores of 70 and above are considered clinical threshold.
8. Variables of the Study

   Dependent Variables of the Study:

   Revised Child Anxiety and Depression Scale - Child Form, Revised Child Anxiety and Depression Scale - Parent Form, Quality of Life Scale for Children.

   Independent Variables of the Study:

   The independent variable of the study was the CBT-based psycho-education program.
9. Data Collection

   The data were collected by face-to-face interviews with children/adolescents diagnosed with ADHD and their parents between September 25, 2023 and August 30, 2024 at Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital/Child and Adolescent Psychiatry Department. A suitable room in the Child and Adolescent Psychiatry Outpatient Clinic was prepared for data collection, and parents were contacted by phone in advance for appointments, and appropriate dates and times were determined.

   Before the data collection started, the child/adolescent diagnosed with ADHD and the family were informed about the study by the specialist/assistant physician working in the Child and Adolescent Psychiatry outpatient clinic who met the inclusion criteria and the contact information of the parents who agreed to participate in the study was recorded. For the sample group, children/adolescents and parents who met the study criteria were ranked in consecutive order by the researcher.

   The sample group, which was determined in consecutive order, was randomly divided into two groups, with odd numbers being the intervention group and even numbers being the control group, and the participants who volunteered to participate in the study were informed about the study and verbal consent was obtained.

   A pre-test was administered to the control group when the first interview was conducted. When they came to the hospital for a follow-up visit 30-40 days later, a post-test was administered. The intervention group was contacted by phone beforehand and the purpose and method of the study was explained again and the date and time for the first interview was determined. A total of 8 sessions were held with the child/adolescent and his/her parent with the individual face-to-face interview technique during the appointment hours determined on weekdays, one session per week. After each session, the date and time of the next session was determined with the parents in the intervention group. Each session lasted 40-45 minutes on average. With the intervention group, a pre-test was administered in the first session and a post-test was administered in the last session. In both groups, data collection tools were filled in by the researcher. This process took 20-25 minutes except for the session time. Anxiety and Depression Scale-Parent Form was filled out based on the mother when both parents were present with the child during the session.
10. Investigative Nursing Initiative

Before starting the study, the researcher completed the training program called "CBT Practitioner Training in Children and Adolescents" (Certificate No: UN_041054323475554869027) from Fatih Sultan Mehmet University Continuing Education Center (Appendix: ). CBT-based psychoeducation booklet prepared by the researcher was used in the sessions.

In the first interview with the children and parents who participated in the study and who were in the intervention group, the first test application (Personal Information Form, Revised Anxiety and Depression Scale-Child/Parent Form and Quality of Life Scale) data were collected. At the doctor's visit 30-40 days later, the post-test was administered. No nursing intervention was applied to the control group other than the pre-test post-test application.

After the first test was performed in the first session with the patients in the intervention group, information about ADHD was given by giving a booklet prepared for parents in the first session (dheb book appendix). Parents were given homework assignments in the psychoeducation booklet prepared for children and adolescents to be included in the sessions themselves and their applications within the session.

ELIGIBILITY:
Inclusion Criteria:

Children who are diagnosed with ADHD according to DSM-V diagnostic criteria,

* Do not have another psychiatric disorder not specific to ADHD,
* Do not have a mental disability,
* Do not seek pharmacological treatment,
* Are between the ages of 8-16,
* Can read and write,
* Can communicate and cooperate,
* Agree to participate in the study (parents and/or themselves) are included in the study.

Exclusion Criteria:

* Those with another psychiatric disorder not specific to ADHD,
* Those with mental retardation,
* Those receiving pharmacological treatment,
* Those between the ages of 8-16,
* Those who cannot read or write,
* Those who request to withdraw from the study

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Psycho-educational application based on Cognitive Behavioral Therapy | 4 weeks
  This study will investigate how cognitive behavior-based psychoeducation given to children diagnosed with Attention Deficit Hyperactivity Disorder will affect the child's quality of life, anxiety, and depression.
  Two scales will be used to measure the results of the interventions made in the research. These scales are:
  1-Child Anxiety and Depression Scale; consists of 47 items.
  2.Quality of life scale for children consists of 23 items.

CONTACTS AND LOCATIONS:
Overall Officials: vedat Argın, lecturer, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital, Kahramanmaraş, OnikiŞubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Argin V, Cigdem Z, Altun H, Doganer A. The effects of cognitive behavioral therapy-based psychoeducation on quality of life, anxiety, and depression in children with attention deficit hyperactivity disorder. BMC Psychol. 2026 Feb 7. doi: 10.1186/s40359-026-04110-7. Online ahead of print. PMID 41652519